CLINICAL TRIAL: NCT04997473
Title: Behavioral Weight Loss Intervention Utilizing Mobile Health Technology in Hematopoietic Stem Cell Transplant Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Theodore Moore, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UCLA BWL001
Record Dates: First submitted 2021-07-23; First posted 2021-08-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Stem Cell Transplant
MeSH Terms: conditions — Obesity | interventions — Telemedicine; Amyloid

STUDY DESIGN:
Intervention Model Description: Evaluate the effectiveness of an addiction model based mobile health (mHealth) weight loss intervention with coaching in obese pediatric patients after hematopoietic stem cell transplant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App Group (Experimental): Participants will be receiving an addiction model based mobile health (mHealth) weight loss intervention with coaching for a total of 4 months duration
  Interventions: Behavioral: W8L2G mobile health (mHealth) app

INTERVENTIONS:
Behavioral: W8L2G mobile health (mHealth) app — Weight loss phone app based on addiction principles. This intervention has been validated in two prior studies. Participants will also interact with coaches throughout the intervention

SUMMARY:
Pilot study enrolling obese post HSCT (hematopoietic stem cell transplantation) patients at the hematology/oncology clinic at the Mattel Children's Hospital, University of California, Los Angeles. Parameters include percent over the 95th percentile (%BMIp95), zBMI, fasting metabolic metrics, addictive eating habits, and motivation for change.

DETAILED DESCRIPTION:
This is a pilot study enrolling obese patients, age 13-30, in an addiction model based smartphone mobile health (mHealth) weight loss intervention with coaching at a minimum of 100 days after hematopoietic stem cell transplantation. Patients will be screened and enrolled by the study coordinator, who will collect/submit biospecimens in addition to patient demographic characteristics and clinical outcomes. At the initial visit and enrollment, equipment will be disbursed to patients along with a schedule that outlines the 4-month intervention plan. After the initial visit, participants will participate in two additional in-clinic visits at 2 months and at the conclusion of the study at 4 months. Participants will also be involved in weekly phone calls and daily weekday texts to discuss their status for the 4 month duration.

This study will then correlate the results in change of BMI with patient characteristics, adherence to intervention, changes in metabolic parameters, physical activity levels, and addictive eating behaviors. Investigators are aiming to recruit a total of 20 adolescents/young adults total. No pilot group is necessary since the feasibility of this intervention has been validated in prior published studies.

The proposed model of delivery makes it possible to: 1) intervene with the participant and provide autonomy, 2) deliver the material over an extended period of time in a more convenient platform for the participant and families, 3) reduce many access barriers common in conventional outpatient obesity interventions, such as transportation or missed days of school and work, and 4) help youth develop skills to overcome their addictive eating behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 13 and ≤ 30 years old with a history of HSCT of any type, at least 100 days post-transplant at initial consultation of the study, will be eligible for the study.
* Both male and female patients will be eligible.
* Patients must classify as obese, represented as Body mass index [BMI] ≥85th percentile for age and gender.
* Patients must also be able to read English since the app intervention is only available in English form.

Exclusion Criteria:

* Patients who are ≤ 13 or ≥ 30 years old are not eligible for the study.
* Patients who are < 100 days post-transplant at initial consultation will not be eligible for the study, but may become eligible if they are >100 days post-transplant at their next consultation that falls within the enrollment window.
* Patients whose BMI does not fall under the obese category will be excluded.
* No patients will be excluded for any specific underlying medical condition, but decisions will be made on a case by case basis if a patient's functioning is deemed to significantly interfere with intervention participation.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2027-01-09 (Estimated); Study Completion 2027-01-09 (Estimated)

PRIMARY OUTCOMES:
BMI | 4 months
  To evaluate the effectiveness of an addiction-based weight loss intervention, embodied as a smartphone app with telephone coaching, on weight (weight and height will be combined to report BMI in kg/m^2) outcomes of overweight and obese post HSCT adolescents and young adults.

SECONDARY OUTCOMES:
Behavioral changes, metabolic parameters, feasibility of app | 4 months
  To evaluate the changes in metabolic parameters and physical activity levels, in addition to modifications in addictive eating behaviors, motivation, and self-regulatory behaviors. To evaluate the feasibility, adherence, and satisfaction of this intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore B Moore, MD, Principal Investigator — UCLA Health
Locations (1):
- UCLA Mattel Children's Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No